CLINICAL TRIAL: NCT03887975
Title: T-Scan Evaluation for Different Types of Occlusion in Mandibular Overdenture Retained By Two Splinted Mini Implants (In Vivo Study)
Brief Title: T-Scan Study of Occlusion in Case of Implant Retained Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Heba tarek abdallah, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ain Shams heba tarek
Record Dates: First submitted 2019-03-09; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Dental Occlusion, Traumatic; Edentulous Alveolar Ridge
MeSH Terms: conditions — Dental Occlusion, Traumatic

STUDY DESIGN:
Intervention Model Description: Completely edentulous patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percentage of force in monoplane occlusion (Active Comparator): Different occlusal scheme evaluation using tscan
  Interventions: Procedure: Monoplane Occlusion
- Percentage of force in lingualized occlusion (Active Comparator): Different occlusal scheme evaluation using tscan
  Interventions: Procedure: Lingualized occlusion

INTERVENTIONS:
Procedure: Monoplane Occlusion — Monoplane and lingualized occlusion effect on force distribution
  Arms: Percentage of force in monoplane occlusion
Procedure: Lingualized occlusion — Monoplane and lingualized occlusion effect on force distribution
  Arms: Percentage of force in lingualized occlusion

SUMMARY:
Materials and methods: fourteen patients were selected according to the inclusion criteria, the participants were stratified equally into two groups, patients were assigned to receive either monoplane or lingualized occlusal schemes to their overdentures. For each patient placement of two mini-implants in the mandible at the canine region was done, bar joint attachment was used to splint the mini implants. Each implant was 2.5 mm in diameter and 10 mm in length. T-scan occlusal load analysis records were done in centric occlusion , the records was used to analyze the biting force of the denture as a Full Closure Force Movie recording, then Time vs. Force Graph of that Force Movie is accomplished. T-scan records were taken three times for each patient in the two groups ,Immediately after loading ,three months and six months of loading.

DETAILED DESCRIPTION:
Fourteen completely edentulous patients will be selected from the outpatient clinic of removable Prosthodontics Department, Faculty of Dentistry, Ain Shams University.

Patient's approval:

All participants were informed in details about the nature of the research and the purpose of the study. They should agree to take part in it and sign an informed consent form.

All reasonable measures to protect the security of the personal information and privacy of the patient protected health information will be taken.

All participants were given notice about their practices and their legal duties and rights.

All participants were informed about their benefits from the research that will be a well-fitting and retentive denture In case of failure of the treatment the patient were informed that a regular complete dentures will be constructed. All data were kept confidential.

Grouping of patients:-

Patients were randomly divided into two equal groups,each group include:

Group (1): seven patients rehabilitated by bar retained mandibular overdenture with lingualized occlusal concept supported by two mini implants.

Group (2): seven patients rehabilitated by bar retained mandibular overdenture with monoplane occlusal concept supported by two mini implants.

Patient examination:

Thorough general and oral examinations were carried out to ensure acceptable conditions for the proposed mini-implant treatment

Oral examination:

Visual and digital examinations were thoroughly carried out to assess the condition of intra-oral tissues and ensure that the patients are suitable for the future surgical and prosthetic procedures.

Construction of complete dentures with lingualized and monoplane occlusal schemes:

For all patients Upper and lower primary impressions were made by using compound impression material . The impression were poured into plaster and acrylic special trays were constructed. Border molding with green stick compound and final impressions for upper and lower ridges were done by using Zinc oxide an eugenol impression material to obtain master casts . Occlusion blocks on the master casts were constructed.

For lingualized group :

face bow record was made to mount the maxillary casts on a semi-adjustable articulator .Centric occluding relation was recorded at the correct occlusal vertical dimension using check bite technique to mount the lower cast on the articulator .

Protrusive record was made to adjust the horizontal condylar guidance of the articulator and the lateral condylar guidance was adjusted according to Hanau's formula (L=H/8+12).

Setting up of the teeth was done using acrylic teeth according to the lingualized concept of occlusion as follow: Anterior teeth were set according to esthetics, phonetics and lip support, Lingual cusps of mandibular posterior teeth were placed medial to the lines drawn from the tip of the canine to both sides of the retromolar pad. The mandibular posterior teeth were placed with no transverse inclination (no Monson curve). The interlocking transverse ridges of the occlusal surface were ground to provide freedom in occlusion (long centric). Maxillary posterior teeth were modified to eliminate buccal cusp contact both in centric and eccentric positions. The upper posterior teeth were arranged with their palatal cusps in the modified central fossae of the lower posterior teeth. In lateral excursions, the posterior teeth were arranged and adjusted to establish bilateral balanced occlusion.

Waxing up of the denture bases was done and try-in was made and the occlusion was carefully checked on the articulator as well as in the patient mouth, the occlusion checked both in centric and eccentric positions.For monoplane group:

Jaw relation was recorded using check bite technique then setting up of the teeth was done according to the monoplane concept of occlusion as follow : Artificial teeth were used after flattening of the cusp inclines. The teeth were arranged anteroposteriorly parallel with the plane of denture foundation. The teeth were arranged mediolaterally with no medial or lateral inclination. The lower second molars were kept out of occlusion. The upper and lower anterior teeth were arranged to establish zero degree incisal guidance.

Waxing up of denture was made and try in was done then occlusion was carefully checked .

for all patients dentures: Flasking, packing and processing were done for waxed up dentures. Laboratory remounting was carried out to correct any occlusal discrepancy from denture processing. Finishing and polishing of the dentures were carried out after their removal from the casts and the dentures were delivered to the patients.

Pre operative cone beam were made to all the patients to Locate the position of mental foramina, identify and measure the anterior loop of mental nerve, measure the inter-foraminal distance and determine the prospective position of mini-implants equi-distant on each side from the midline by using clear acrylic surgical stent duplicated from the lower denture with gutta percha attached to the proposed implant sites.

patients were instructed to take the following pre-surgical medications: Antibiotic (Clavulanate-Potentiated Amoxycillin 1gm) every 12 hours started the day before surgery and continued for one week, Analgesic and anti-inflammatory drug (Diclofenac Sodium 50mg) every 8 hours started 1 hour before surgery and continued for one week, Mouth wash (Chlorohexidine Gluconate ) every 8 hours started the day before surgery and continued for one week. Patients were instructed to rinse with Chlorohexidine Gluconate mouth wash at the time of the operation. Bilateral mandibular nerve block (Articaine Hydrochloride 4% with Epinephrine 1:100,000) was administrated, with infiltration anesthesia at the surgical field.

The Surgical stent was used to guide the insertion of the two mini implants in the anterior area between the two mental foramina, where a probe was entered in each hole and piercing the mucosa leaving a bleeding points.

At the marked implant site, tissue punch was used to remove the soft tissue prior to the use of the pilot drill . A 1.3 mm pilot drill was lightly pumped up and down vertically perpendicular to the occlusal plane through the holes of the surgical stent, penetrating the crestal bone 3-4 mm.

Sterile internal and external saline irrigation was used throughout the drilling procedure. The pilot holes were deepened to a depth of the implants to be placed using osteotomy drill of 10 mm. The MDI vial was opened and the mini implant 2.5mm diameter, 10mm length was carried to the osteotomy site, and was rotated in a clockwise direction while exerting a slight downward pressure using a finger rachet driver. The wrench torque was connected to rachet driver (with the directional arrow facing a clockwise).

The final stage of the MDI placement was carried out with a careful controlled turns for complete seating, 1/4 turn rotation with 15 seconds pauses between rotations Mini-implant placement was completed with the protrusion of the full length of the abutment head from the mucosa, but with no thread portions visible.

The square head of implants trimmed to the first mark that allow fixed abutment heights suitable for the available inter arch space for all patients groups.

Bar attachment construction:

Closed tray impression was made with rubber base putty impression material using plastic Transfer coping and implant analogue. Stone was poured to get cast with implant analogue in its place representing patient's mouth. Metal custom made bar constructed splinting the two mini implants.

Bar cemented with self adhesive resin cement "G-Cem capsule" and excess removed around the bar and mucosa. A fast-setting chair side Poly-vinyl siloxane material (PVS) was loaded onto the fitting surface of the lower denture , then it was seated in the patient's mouth to locate the position of the bar, after few minutes the denture was removed from the patient's mouth and area marked by the bar removed using large round bur. The denture was inserted in the patient's mouth to ensure that it was passively seated.

Small amount of putty PVS used to block under and around the bar for pick up procedure .Clip seated in it's place and Auto-polymerizing acrylic resin in dough stage was applied in the space created in the denture opposite to the bar clip, and the overdenture was seated on the model. Firm steady pressure was applied on the overdenture bilaterally till complete curing of the resin. The excess material was trimmed and smoothened.

T-scan occlusal stress distribution recording:

T-Scan device was used, the Device consists of:

Scan handle and lab-top. Box of large and box of small sensors. Box of large and box of small sensor supports. The sensor support provided enough width to cover the molars and the patients were allowed to close comfortably, tried in to choose the correct support size.

sensors support was attached to the T-Scan handle with the "Sensor Position Guide" faced up until it clicks into place. The latch was lifted and the sensor was inserted, which were the same size as support, so that the outside edges of the sensor slide into the sensor support channels then the latch was closed to lock the center in place.

A green light indicated that the sensor was properly connected.

Patient Record:

Records done in centric position by the following steps:

Patient record was created by clicking "New Patient", and the patient information, first, middle and last name, gender, date of birth and ID number was filled.

The sensor was inserted into the mouth like that in impression tray. Patient opened his/her mouth slightly. The sensor was inserted so that the position guide touch the central incisor at the mid line. The sensor was held in place so that the sensor level with the occlusal plane.

T-Scan device show range of colors to differentiate the forces on the teeth, Adjusting sensitivity to ensure the entire color spectrum is used to visualize the differences in these forces and that the maximum forces are within the sensor forces range, and this was done by:

* The patients were asked to bit and clench firmly. The patients were asked to clench and the tooth contact was observed on the screen. The ideal setting is maximum 3 pink contact.
* Records taken at centric positions

Rechecking occlusion and occlusal load equilibration in patients mouth:

Patients were frequently recalled for inspection, post insertion adjustments, future denture relining and T-scan measurements done to assess occlusal forces immediately after loading, at 3 and 6 months after loading.

After three months of loading patients of lingualized group complained from denture movement in the posterior region.

Chair side soft liner was added to the fitting surface of the dentures to adjust the posterior occlusion and to comfort the patients. They were guided to close in centric position till the soft liner material set . The occlusal equilibration were checked and t-scan records made to measure occlusal stresses distribution.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 50-65. Free from any systemic diseases affecting bone metabolism.
* Free from tempromandibular joint disorders.
* Having normal ridge relationship.
* Adequate interarch space.
* No parafunctional habits.
* Residual ridge with adequate height covered by firm dense fibrous mucoperiosteum with no sharp spicules.

Exclusion Criteria:

* systemic diseases affecting metabolism of bone e.g bone diseases, hyperparathyroidism and renal diseases
* Severe blood disease (hemophilia ect)
* Severe vascular heart disease
* Liver problems
* Severe immunodeficiency .Patients who are undergoing strong chemotherapy,Irradiated patients or requiring hard or soft tissue grafting of the proposed implant site.
* Uncooperative patients who have no understanding of the need for regular follow-up .Patient diagnosed with neuromuscular disorders, para functional habits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
traumatic dental occlusion by T-Scan III | 6months
  To evaluate the stress distribution in mandibular overdenture retained by two splinted mini implants using monoplane and lingualized occlusion in setting of teeth using T-Scan.

CONTACTS AND LOCATIONS:
Overall Officials: Heba T Mohamed, Doctor, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No